CLINICAL TRIAL: NCT00004767
Title: Phase II Study of Sodium Phenylbutyrate, Sodium Benzoate, Sodium Phenylacetate, and Dietary Intervention for Urea Cycle Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11753; JHUSM-11753
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Amino Acid Metabolism, Inborn Errors
Keywords: inborn errors of metabolism; rare disease; urea cycle disorder
MeSH Terms: conditions — Amino Acid Metabolism, Inborn Errors; Metabolism, Inborn Errors; Rare Diseases; Urea Cycle Disorders, Inborn | interventions — Sodium Benzoate; phenylacetic acid; 4-phenylbutyric acid; Diet Therapy

INTERVENTIONS:
Drug: Sodium Benzoate
Drug: Sodium Phenylacetate
Drug: Sodium Phenylbutyrate
Behavioral: Dietary Intervention

SUMMARY:
OBJECTIVES:

I. Assess the safety and efficacy of sodium phenylbutyrate, sodium benzoate, sodium phenylacetate, and dietary intervention in patients with urea cycle disorders.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This protocol describes several clinical studies of pharmacologic and dietary management in patients with urea cycle disorders.

Patients with carbamyl phosphate synthetase and ornithine transcarbamylase deficiency are treated with a low-protein diet, essential amino acids (for neonatal onset disease), caloric supplementation, oral sodium phenylbutyrate (now approved as a prescription drug 11/97), and citrulline or arginine free base.

Patients with argininosuccinic acid synthetase deficiency are treated with a low-protein diet, caloric supplementation, oral sodium phenylbutyrate (now approved as a prescription drug 11/97), and arginine free base.

Patients with argininosuccinic aciduria (AA) are treated with a low-protein diet, caloric supplementation, and arginine free base. (Discontinued 11/97) Any patient who develops hyperammonemia is treated with intravenous sodium benzoate, sodium phenylbutyrate, and arginine hydrochloride; benzoate and phenylbutyrate are not given to patients with AA.

If ammonium stabilizes at normal or near normal levels, intravenous medications are gradually replaced by oral medications. If there is no significant decrease in ammonium within 8 hours, patients begin hemodialysis.

Concurrent therapy with ondansetron, high caloric intake, and mannitol for elevated intracranial pressure is allowed. Dietary and intravenous nitrogen is prohibited. (Discontinued 11/97)

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Urea cycle deficiency, i.e.: Carbamyl phosphate synthetase deficiency (CPSD) Ornithine transcarbamylase deficiency (OTCD) Argininosuccinic acid synthetase deficiency (ASD) Argininosuccinic aciduria (AA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1985-01

CONTACTS AND LOCATIONS:
Overall Officials: Saul W. Brusilow, Study Chair — Johns Hopkins University